CLINICAL TRIAL: NCT06574451
Title: Effectiveness and Safety of Adjuvant Software Based on Virtual Reality for Post-thoracoscopic Surgery Pain (VR-TSP)
Brief Title: Effectiveness and Safety of Adjuvant Software Based on Virtual Reality for Post-thoracoscopic Surgery Pain
Acronym: VR-TSP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Guang Dong Liang Zi Health Consulting Co., Ltd, Guang Dong, China. (Unknown); Tianjin Medical University General Hospital (Other); Ruijin Hospital (Other); Maoming People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VR-TSP
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-04

CONDITIONS: Acute Postoperative Pain; Video-assisted Thoracic Surgery; Virtual Reality
Keywords: Acute Postoperative Pain; VATS; VR
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-assisted postoperative analgesia group (Experimental): Patients will receive postoperative analgesic adjunctive therapy software to assist in pain control, with one postoperative analgesic adjunctive therapy software intervention at 24 hours and 48 hours after surgery, and pain evaluation within 30 minutes.
  All participants will receive intravenous analgesics pumped with mechanical pumps (analgesic pumps: Flurbiprofen cilexil Injection 5ml: 50mg/stick*4 sticks, combined with Dezocine Injection 1ml: 5mg/stick*6 sticks, add Ondansetron Hydrochloride Injection: 2ml: 4mg/stick*2 sticks; or add Tolisetron Mesylate Injection: 2ml: 6 mg/stick*4 sticks, diluted to 100mL with 0.9% sodium chloride injection).In case of an outbreak of pain (when analgesic pump is ineffective and the pain is unbearable), analgesic medication regimen: flurbiprofen cilofen injection 5 ml: 50 mg/piece, intravenous injection.
  Interventions: Device: VR-assisted postoperative analgesia
- Non-VR-assisted analgesia group (No Intervention): The control group will not experience postoperative analgesic adjuvant therapy software and will only record the pain level within 30 minutes at 24 hours and 48 hours after surgery.
  All participants will receive intravenous analgesics pumped with mechanical pumps (analgesic pumps: Flurbiprofen cilexil Injection 5ml: 50mg/stick*4 sticks, combined with Dezocine Injection 1ml: 5mg/stick*6 sticks, add Ondansetron Hydrochloride Injection: 2ml: 4mg/stick*2 sticks; or add Tolisetron Mesylate Injection: 2ml: 6 mg/stick*4 sticks, diluted to 100mL with 0.9% sodium chloride injection).In case of an outbreak of pain (when analgesic pump is ineffective and the pain is unbearable), analgesic medication regimen: flurbiprofen cilofen injection 5 ml: 50 mg/piece, intravenous injection.

INTERVENTIONS:
Device: VR-assisted postoperative analgesia — Patients will receive postoperative analgesic adjunctive therapy software to assist in pain control, with one postoperative analgesic adjunctive therapy software intervention at 24 hours and 48 hours after surgery, and pain evaluation within 30 minutes.
  Arms: VR-assisted postoperative analgesia group

SUMMARY:
A randomized controlled, prospective, multicenter, open label, superiority trial aims to evaluate the effectiveness and safety of adjuvant software based on virtual reality for post-thoracoscopic surgery pain.

DETAILED DESCRIPTION:
215 eligible patients will be enrolled. All enrolled patients will have an NRS score at 24 hours postoperatively, and those with a score greater than or equal to 4 will be randomly assigned to the test and control groups.

Patients in the experimental group will receive postoperative analgesic adjunctive therapy software to assist in pain control, with one postoperative analgesic adjunctive therapy software intervention at 24 hours and 48 hours after surgery, and pain evaluation within 30 minutes.

The control group will not experience postoperative analgesic adjuvant therapy software and will only record the pain level within 30 minutes. Subjects will complete a study summary form upon completion of follow-up.

All participants will receive intravenous analgesics pumped with mechanical pumps (analgesic pumps: Flurbiprofen cilexil Injection 5ml: 50mg/stick*4 sticks, combined with Dezocine Injection 1ml: 5mg/stick*6 sticks, add Ondansetron Hydrochloride Injection: 2ml: 4mg/stick*2 sticks; or add Tolisetron Mesylate Injection: 2ml: 6 mg/stick*4 sticks, diluted to 100mL with 0.9% sodium chloride injection).In case of an outbreak of pain (when analgesic pump is ineffective and the pain is unbearable), analgesic medication regimen: flurbiprofen cilofen injection (5 ml): 50 mg/piece, intravenous injection.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age greater than or equal to 18 years.

  2.Patients within 1 day after thoracoscopic surgery.

  3.Junior high school degree or above, Mandarin communication is unimpeded, with certain Internet knowledge and mobile phone reading and writing skills.

  4.The score of the numeric grading scale (NRS) at 24 hours postoperatively ≥ 4 points.

  5.Patients who are able to understand the purpose of the study, voluntarily participate in and sign the informed consent form, and are willing to complete the follow-up as required by the protocol.

Exclusion Criteria:

* 1.Patients with severe cognitive impairment.

  2.Patients with a previous diagnosis of epilepsy, dementia, migraine, or other neurological disease that may result in the inability to use postoperative analgesic adjuvant therapy software or that may have adverse effects.

  3.Patients who are unable to understand or speak Mandarin.

  4.Patients who have visual abnormalities, severe hearing impairment, or motion sickness, etc., and are unable to view VR.

  5.Patients with trauma to the eyes, face, or neck that prevents the comfortable use of the VR device.

  6.Patients with severe heart, liver, kidney, hematologic, digestive, nervous system diseases and malnutrition.

  7.Patients who have previously used virtual reality software for pain that has not responded to treatment.

  8.Patients with a history of severe alcohol abuse, long-term heavy drinking, and symptoms of alcohol dependence.

  9.Patients who have participated in any analgesic interventional study within the past 1 week.

  10.Females who are pregnant or plan to become pregnant during the study.

  11.The patient or their immediate family member works for a digital health or pharmaceutical company for acute or chronic pain treatment.

  12.Patients who are unable to use electronic devices such as smartphones.

  13.Other conditions that the investigator considers inappropriate for participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2023-04-22 (Actual); Primary Completion 2025-04-24 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | The NRS evaluation is within 30 minutes of 24 and 48 hours after surgery.
  The NRS score is a commonly used postoperative pain assessment tool. The score uses a numeric scale from 0 to 10, on which patients are asked to mark their level of pain, with 0 being no pain and 10 being the most severe pain.

SECONDARY OUTCOMES:
Incidence of adverse events | Assessment of adverse events is completed within 2 days postoperatively
  Any unfavorable medical occurrence during the course of the study, whether device-related or not, is an adverse event.
Incidence of serious adverse events | Assessment of serious adverse events is completed within 2 days postoperatively
  If an event occurs during the clinical study that results in death or serious deterioration of health status, it is judged to be a serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Zhao Zhong, Principal Investigator — Guangdong Provincial People's Hospital
Locations (4):
- China (4):
  - Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong
  - Maoming People's Hospital, Maoming, Guangdong
  - Ruijing Hospital, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality